CLINICAL TRIAL: NCT06557512
Title: A Pilot Trial of Adjuvant Hypofractionated Stereotactic Radiosurgery for Intermediate-risk Meningioma (SRS-AIM)
Brief Title: Adjuvant Hypofractionated Stereotactic Radiosurgery for Intermediate-risk Meningioma
Acronym: SRS-AIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24724; NCI-2024-06542 (Registry Identifier: NCI Clinical Trials Reporting Program (NCI CTRP))
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Meningioma; Meningioma, Malignant; Recurrent Meningioma
MeSH Terms: conditions — Meningioma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hypofractionated Stereotactic Radiosurgery (SRS) (Experimental): Participants undergo hypofractionated stereotactic radiosurgery over 15-30 minutes QD on days 1-5 in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Hypofractionated Stereotactic Radiosurgery (SRS); Procedure: Magnetic Resonance Imaging (MRI); Procedure: Computed Tomography (CT)

INTERVENTIONS:
Radiation: Hypofractionated Stereotactic Radiosurgery (SRS) — Undergo Hypofractionated Stereotactic Radiosurgery
  Other Names: Fractionated Stereotactic Radiation Therapy; SRS
Procedure: Magnetic Resonance Imaging (MRI) — Undergo MRI
  Other Names: MRI; MR
Procedure: Computed Tomography (CT) — Undergo CT imaging
  Other Names: CT

SUMMARY:
This clinical trial tests the safety and effectiveness of hypofractionated stereotactic radiosurgery for treating patients who have undergone surgical resection for grade II meningiomas or grade I meningiomas that have come back after a period of improvement (recurrent). Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill tumor cells and shrink tumors. Stereotactic radiosurgery is a type of external radiation therapy that uses special equipment to position a patient and precisely deliver radiation to tumors in the body. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Hypofractionated stereotactic radiosurgery may be safe, tolerable, and effective in treating patients with grade II or recurrent grade I meningiomas after surgical resection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety of adjuvant hypofractionated stereotactic radiosurgery after gross total resection of intermediate risk meningioma.

SECONDARY OBJECTIVES:

I. To report the efficacy of adjuvant hypofractionated stereotactic radiosurgery in participants with intermediate risk meningioma.

II. To evaluate the 3-year overall survival rate of participants treated with adjuvant stereotactic radiosurgery.

III. To report on the financial impact, quality of life, and treatment burden of participants who undergo adjuvant stereotactic radiosurgery.

EXPLORATORY OBJECTIVES:

I. To prospectively collect and assess a prognostic and predictive gene expression panel biomarker and deoxyribonucleic acid (DNA) methylation based genomic classification systems for meningioma.

II. To report the comparative dosimetry of adjuvant stereotactic radiosurgery as compared to simulated external beam plans generated based on the drawn planning target volumes.

OUTLINE:

Participants undergo hypofractionated stereotactic radiosurgery over 15-30 minutes once daily (QD) on days 1-5 in the absence of disease progression or unacceptable toxicity. Additionally, participants undergo magnetic resonance imaging (MRI) throughout the study and may undergo computed tomography (CT) as necessary.

After completion of study treatment, participants are followed up at months 3 and 6 and then at years 1, 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Age >+ 18 years at time of study entry
* Ability to understand and the willingness to sign a written informed consent document.
* Histologic diagnosis of newly diagnosed World Health Organization (WHO) grade 2 or recurrent WHO grade 1 meningioma. With regard to recurrent WHO grade 1 meningioma, participants must present with radiographic evidence of recurrence, and have a histologic diagnosis of WHO grade 1 meningioma at the most recent resection.

  * Note: For participants diagnosed outside of University of California San Francisco (UCSF), re-review of pathology at UCSF is strongly encouraged. Hematoxylin and eosin (H&E) slides will be reviewed by UCSF pathologists.
* Participants must have undergone a gross-total surgical resection as deemed by their neurosurgeon (Simpson grade I-III resection), using all available information which can include post-operative MRI, of a meningioma within 180 days of enrollment.
* Participants must have a pre-operative MRI.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Karnofsky score of 70 or higher)
* Participants must have post-operative MRI indicating anatomy suitable for hypofractionated radiosurgery, as reviewed by the Radiation Oncology co-principal investigators (PIs).

Exclusion Criteria:

* Concurrent participation in another clinical study with an investigational product unless it is an observational (non-interventional) study or the follow-up period of an interventional study.
* Extensive multifocal (3 or more meningiomas) or metastatic disease.
* Participants with tumors within 2mm of the optic apparatus or brainstem will be excluded.
* Participants with another active primary malignancy or history of previous malignancy (except non-melanoma skin cancers, low and favourable-intermediate risk prostate cancers, and in situ cancers such as bladder, gastric, colon, cervical/dysplasia, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry and no additional therapy is required or anticipated to be required during the study period.
* Female participants who are pregnant.
* Any underlying medical or psychiatric condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of participant safety or study results.
* Participants with uncontrolled seizures, defined as greater than 3 disabling seizures per day while on anti-epileptic drugs.
* Participants who have had previous intracranial radiotherapy overlapping with the area that would be targeted for stereotactic radiosurgery by this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with reported adverse events | Up to 1 year
  Adverse events will be classified and graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The proportion of CTCAE grade 3-5 toxicity within 1 year of radiation will be estimated along with the exact 90% confidence interval.

SECONDARY OUTCOMES:
Median Local Freedom from recurrence (LFFR) | Up to 3 years
  Local freedom from recurrence (LFFR) is defined as time from start of treatment to date of an event as defined by the above criteria, dated to the imaging study date on which recurrence was assessed. The 3-year LFFR will be estimated by the Kaplan-Meier method. Median LFFR will be estimated, if possible, from the Kaplan-Meier method.
Median Progression-Free Survival (PFS) | Up to 3 years
  Progression free survival (PFS) is defined as the duration of time from start of treatment to date of death or progressive disease (PD) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, dated to the imaging study date on which PD was assessed. The 3-year PFS will be estimated by the Kaplan-Meier method. Median PFS will be estimated, if possible, from the Kaplan-Meier method.
Median overall survival (OS) | Up to 3 years
  Overall survival (OS) is defined as the duration of time from start of treatment to date of death or censored at the date of final visit if lost to follow-up. The 3-year OS will be estimated by the Kaplan-Meier method. Median OS will be estimated, if possible, from the Kaplan-Meier method.
Mean score on the Comprehensive Score for Financial Toxicity-Functional Assessment of Chronic Illness Therapy (COST-FACIT) over time | Up to 3 months
  The COST-FACIT is an 11-item measure used to assess financial toxicity. Each item is measured on a five-point Likert scale (0 = not at all, 4 = very much), with recall based on the past 7 days related to the participant's disease management. A score is computed by first reverse coding seven items, then taking the sum of all items, multiplying the sum by 1the number of items on the scale, and dividing that number by the number of items answered. Higher scores indicate better Financial Well-Being.
Frequency of responses on the Brief Work and Transportation Survey | Up to 3 months
  The Brief Work and Transportation Survey contains 10-items modeled after items from the National Health Interview Survey asking participants information about current employment, time taken off work for cancer treatment, the transportation burden, and time burden of treatment). Items will be reported categorically based on most frequent response.
Mean score Decision Regret Scale (DRS) | Up to 1 year
  The 5-item Decision Regret Scale was developed to measure regret after health-care decisions Item responses are scored on a scale from 1 (strongly agree) to 5 (strongly disagree). Two of the items are reverse coded and total scores are transformed to a scale of 0-100 by subtracting 1 from each item then multiply the response by 25. To obtain a final score the items are summed and averaged. A score of 0 means no regret and a score of 100 indicates very high regret.
Mean score on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) 30 - Global Health Status over time | Up to 3 years
  The global health status score consists of responses to two items with responses ranging from 1="very poor" to 4="excellent". The raw score is calculated by estimating the mean of the two items that make up the global health scale with a resulting total range of 1-7. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score for the global health status represents a higher quality of life.
Mean score on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) 30 - Functional Domains over time | Up to 3 years
  The functional domains measure the quality of life in Physical functioning, Role functioning, Emotional functioning, Cognitive functioning, Social functioning. Scores consists of responses to items with responses ranging from 1="Not at all" to 4="Very Much". The raw score is calculated by estimating the mean of the items that make up each domains with a resulting total range of 1 - 4. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score for the functional domains represents a high level of functioning
Mean score on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) 30 - Symptoms over time | Up to 3 years
  The Pain score consists of responses to two items with responses ranging from 1="Not at all" to 4="Very Much". The raw score is calculated by estimating the mean of the two items that make up the pain scale with a resulting total range of 1-4. These scores are then transformed to standardized scale score, so that scores range from 0 to 100. A high score for the pain scale / item represents a high level of symptomatology / problems.
Mean score on the EORTC QLQ Brain Cancer Module (BN20) over time | Up to 3 years
  The EORTC QLQ-BN20 consists of 20 questions; seven single item symptom scales (headaches, seizures, drowsiness, hair loss, itchy skin, leg weakness and bladder control), along with four multi-item scales (future uncertainty, visual disorder, motor dysfunction and communication deficit). Raw scores for the QLQ-BN20 items are computed by calculating the mean of the items in each subscale, or the item for each individual and linearly transform the scores to a 0-100 scale. A higher score represents worse QOL for all QLQ-BN20 scales and single items.

CONTACTS AND LOCATIONS:
Overall Officials: William Chen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No